CLINICAL TRIAL: NCT04025151
Title: Nurse-led Alcohol Brief Intervention Plus Mobile Personalized Chat-based Support on Reducing Alcohol Use in University Students: a Pragmatic Randomized Controlled Trial
Brief Title: Nurse-led Alcohol Brief Intervention Plus Mobile Personalized Chat-based Support on Reducing Alcohol Use in University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chat-based ABI (UniStudents)
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Misuse
Keywords: chat-based IM; alcohol brief intervention; alcohol misuse; university students
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Alcohol brief intervention, leaflets, regular personalized messages on ABI through IM Apps, real-time chat-based support through IM Apps
  Interventions: Behavioral: Alcohol brief intervention; Behavioral: 12-page health warning leaflet; Behavioral: Regular messages through Instant Messaging (IM); Behavioral: Real-time chat-based support through IM Apps; Behavioral: AUDIT score interpretation sheet adapted from the Department of Health of Hong Kong
- control group (Active Comparator): Alcohol brief intervention, leaflets, regular messages on general health through SMS
  Interventions: Behavioral: Alcohol brief intervention; Behavioral: 12-page health warning leaflet; Behavioral: General health through SMS; Behavioral: AUDIT score interpretation sheet adapted from the Department of Health of Hong Kong

INTERVENTIONS:
Behavioral: Alcohol brief intervention — At baseline, subjects will receive face-to-face or online alcohol brief intervention developed based on the guideline by the World Health Organisation in 5-10 minutes
Behavioral: 12-page health warning leaflet — Nurses will provide information about the consequences of drinking using a 12-page health warning booklet. Benefits of reducing and quit drinking will be emphasized by focusing on improving their perception towards the impacts on health, social problems, risky behaviors, academic performance and financial issues.
Behavioral: Regular messages through Instant Messaging (IM) — A total of 26 e-messages will be scheduled: once daily for the first week, 3 time/week for subsequent 4 weeks and 1 time/week for the remaining 7 weeks. The frequency will be adjusted according to IM Apps conversation and subject's requests.
  Arms: Intervention group
Behavioral: Real-time chat-based support through IM Apps — The chat-based IM support is the extension of baseline ABI and regular e-messages, which aims to provide real-time behavioral and psychosocial support to reduce or quit drinking. It will be personalized according to the subjects' characteristics (gender, drinking pattern and alcoholic drinks preferences), intention to drink and specific questions regarding drinking. Through real-time chatting (text and/or voice), drinkers can acquire information on consequences of drinking and gain social support immediately to reduce intention to drink and alcohol consumption.
  Arms: Intervention group
Behavioral: General health through SMS — After baseline, they will receive regular e-message through SMS with similar frequency to Intervention group with content on general health and the reminding the importance of participating in the follow-up surveys.
  Arms: control group
Behavioral: AUDIT score interpretation sheet adapted from the Department of Health of Hong Kong — a diagram explaining drinking behaviour and potential health risks, definitions of "alcohol unit" and "binge drinking", and advise on limiting daily drinking to 2 alcohol units for men and 1 unit for women

SUMMARY:
This study aims to assess the effect of personalized support using instant messaging application on alcohol drinking reduction in university students proactively recruited from universities in Hong Kong.

DETAILED DESCRIPTION:
The government has promoted Hong Kong as the Asian's wine hub with zero alcohol tax (ethanol ≤30%) since 2008, which causes dramatic increases in alcohol drinking and binge drinking rates. Alcohol use in youth is the leading cause of disability adjusted life-years loss. Most adult drinkers start drinking at age 18-21. Evidence shows that alcohol brief intervention (ABI) is effective reducing hazardous and harmful alcohol use in university students. The proposed trial aims to enhance the ABI by incorporating information communication technologies (ICTs) such as instant messaging (IM) Apps (e.g. WhatsApp and WeChat) to provide personalized, real-time chat-based support led by nurses. The aims of study are as follows:

1. To determine the main effect of the Intervention vs. Control group on alcohol consumption per week at 6-month (Primary)
2. To assess the effects on alcohol consumption per week at 12-month, AUDIT scores at 6 and 12-month, perceived usefulness of IM app at 12-month, intention to use IM app to reduce/quit drinking at 12-month, number of standard drinks, episode of binge drinking, episode of heavy drinking, planned drinking, Academic Role Expectation and Alcohol Scale, Alcohol Problems Scale, Patient Health Questionnaire 4-item, Perceived Stress Scale 4-item, Covid-19 related drinking behavioral changes, and self-efficacy to reduce/quit drinking at 6-month and 12-month
3. To identify mediators between intervention and outcomes to inform the potential mechanisms
4. To qualitatively explore experience on the interventions for reducing alcohol use and related harms

ELIGIBILITY:
Inclusion Criteria:

* Student aged ≥18 years from local universities in Hong Kong
* Able to read and communicate in Chinese (Cantonese or Mandarin)
* Likely to stay in Hong Kong for most of the time in the next 12 months
* Using IM Apps (WhatsApp or WeChat) installed on a smartphone
* Baseline AUDIT screening score ≥8

Exclusion Criteria:

* Having a history of psychiatric/psychological disease or currently on regular psychotropic medications
* Currently participating in treatments or programmes on reducing alcohol use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Amount of alcohol consumption per week (gram/week) at 6-month follow-up | 6-month after baseline
  Assessed by unit in gram and compare the alcohol consumption between intervention and control group at 6-month after baseline.
Compare the primary outcome using intention-to-treat (ITT), per-protocol (PP) and as-treated (AP) analysis with Compliance Average Causal Effect (CACE) analysis | 6-month after baseline
  To estimate large, moderate and null (same as the control) treatment effects and check whether ITT, AP and PP analysis estimates are biased compared with CACE estimates (alcohol consumption per week at 6-month follow-up)

SECONDARY OUTCOMES:
Amount of alcohol consumption per week (gram/week) at 12-month follow-up | 12-month after baseline
  Assessed by unit in gram and compare the alcohol consumption between intervention and control group at 12-month after baseline.
AUDIT scores at 6-month follow-up | 6-month after baseline
  Assessed by Alcohol Use Disorders Identification Test (ranged 0-40 with higher score indicating problematic alcohol use) and compare the AUDIT between intervention and control group at 6-month after baseline.
AUDIT scores at 12-month follow-up | 12-month after baseline
  Assessed by Alcohol Use Disorders Identification Test (ranged 0-40 with higher score indicating problematic alcohol use) and compare the AUDIT between intervention and control group at 12-month after baseline.
Number of standard drinks (10g of alcohol) per week at 6-month follow-up | 6-month after baseline
  Assessed by either increase or decrease in standard drinks number and compared between intervention and control group at 6-month
Number of standard drinks (10g of alcohol) per week at 12-month follow-up | 12-month after baseline
  Assessed by either increase or decrease in standard drinks number and compared between intervention and control group at 12-month
Episode of binge drinking in the past 30-day at 6-month follow up | at 6-month after baseline
  Defined by 5 standard drink [male] or 4 standard drink [female] in one occasion for binge drinking and compare the episode of binge drinking between intervention group and control at baseline and 6-month follow-up questionnaires
Episode of binge drinking in the past 30-day at 12-month follow up | at 12-month after baseline
  Defined by 5 standard drink [male] or 4 standard drink [female] in one occasion for binge drinking and compare the episode of binge drinking between intervention group and control at baseline and 12-month follow-up questionnaires
Episode of heavy drinking in the past 30-day at 6-month follow up | at 6 -month after baseline
  Defined by 15 standard drink [male] or 8 standard drink[female] in a week for heavy drinking and compare the episode of heavy drinking between intervention group and control at baseline and 6-month follow-up questionnaires
Episode of heavy drinking in the past 30-day at 12-month follow up | at 12-month after baseline
  Defined by 15 standard drink [male] or 8 standard drink [female] in a week for heavy drinking and compare the episode of heavy drinking between intervention group and control at baseline and 12-month follow-up questionnaires
Planned drinking measured in the coming 30-day at 6-month follow up | at 6-month after baseline
  Compare the number of planned drinking (yes or no) between intervention group and control group at baseline and 6-month follow-up questionnaires
Planned drinking measured in the coming 30-day at 12-month follow up | at 12-month after baseline
  Compare the number of planned drinking (yes or no) between intervention group and control group at baseline and 12-month follow-up questionnaires
Academic Role Expectation and Alcohol Scale at 6-month follow-up | at 6-month after baseline
  The four items in this scale addressed the number of times the student had been 'late to class', 'missed class', was 'unable to concentrate' and 'failed to complete assignment' (score range 0-16). The responses included 'not at all', 'once', 'twice', 'three times' and 'four times or more'. The score will be compared between intervention group and control group at baseline and 6-month follow-up questionnaires
Academic Role Expectation and Alcohol Scale at 12-month follow-up | at 12-month after baseline
  The four items in this scale addressed the number of times the student had been 'late to class', 'missed class', was 'unable to concentrate' and 'failed to complete assignment' (score range 0-16). The responses included 'not at all', 'once', 'twice', 'three times' and 'four times or more'. The score will be compared between intervention group and control group at baseline and 12-month follow-up questionnaires
Alcohol Problems Scale at 6-month follow-up | at 6-month after baseline
  The 14-item measure of alcohol-related personal, social, sexual, and legal problems (eg, being physically aggressive toward someone while under the influence of alcohol).The score will be compared between intervention group and control group at baseline and 6-month follow-up questionnaires
Alcohol Problems Scale at 12-month follow-up | at 12- month after baseline
  The 14-item measure of alcohol-related personal, social, sexual, and legal problems (eg, being physically aggressive toward someone while under the influence of alcohol).The score will be compared between intervention group and control group at baseline and 12-month follow-up questionnaires
Mediation analysis of variables at 6-month on weekly amount of alcohol consumption at 12-month | at 12- month after baseline
  Mediation analysis of 6-month factors (knowledge of alcohol drinking, perception of alcohol drinking, intention to quit drinking, mental health) on weekly amount of alcohol consumption at 12-month
Subgroup analysis of baseline intention to quit/reduce drinking | at 12- month after baseline
  Subgroup analysis to check whether the intervention is more effective with participants with intention to quit/reduce drinking on outcomes
Content analysis of IM Apps conversation using alcohol BCT taxonomy | at 12- month after baseline
  The conversations between the participants and the nurse will be analyzed and categorized into different sub-type of BCT taxonomy
Patient Health Questionnaire 4-item (PHQ-4) at 6-month | at 6-month after baseline
  Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression. The score will be compared between intervention group and control group at baseline and 6-month follow-up questionnaires
Patient Health Questionnaire 4-item (PHQ-4) at 12-month | at 12-month after baseline
  Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression. The score will be compared between intervention group and control group at baseline and 12-month follow-up questionnaires
Perceived Stress Scale 4-item (PSS-4) at 6-month | at 6-month after baseline
  Subjects' responses are measured on a five-point scale (0 = never, 1 = almost never, 2
  =sometimes, 3 = fairly often, 4 = very often). Scoring: PSS-4 scores are obtained by summing across all four items. Scoring items 2 and 3 require reverse coding. This involves assigning the opposite score. For example, a score of 0=4, 1=3, 2=2, 3=1, and 4=0. The higher the score, the more perceived stress.
  The score will be compared between intervention group and control group at baseline and 6-month follow-up questionnaires
Perceived Stress Scale 4-item (PSS-4) at 12-month | at 12-month after baseline
  Subjects' responses are measured on a five-point scale (0 = never, 1 = almost never, 2
  =sometimes, 3 = fairly often, 4 = very often). Scoring: PSS-4 scores are obtained by summing across all four items. Scoring items 2 and 3 require reverse coding. This involves assigning the opposite score. For example, a score of 0=4, 1=3, 2=2, 3=1, and 4=0. The higher the score, the more perceived stress.
  The score will be compared between intervention group and control group at baseline and 12-month follow-up questionnaires
Perceived usefulness of IM app intervention at 12-month | at 12-month after baseline
  Score ranges from 0 to 10 with higher score indicates a higher level of usefulness of our intervention.
Intention to continue using IM app intervention at 12-month | at 12-month after baseline
  Ask for intention to use (yes/no) IM app intervention to reduce/quit drinking at 12-month
Self-efficacy to reduce/quit drinking at 6-month | at 6-month after baseline
  Perceived difficulty, confidence and importance of quitting/reducing to drink will be asked.
  Score ranges from 0 to 10 with higher score indicates a high level. The score will be compared between intervention group and control group at baseline and 6-month follow-up questionnaires
Self-efficacy to reduce/quit drinking at 12-month | at 12-month after baseline
  Perceived difficulty, confidence and importance of quitting/reducing to drink will be asked.
  Score ranges from 0 to 10 with higher score indicates a high level. The score will be compared between intervention group and control group at baseline and 12-month follow-up questionnaires
Covid-19 related drinking behavioral changes at baseline | at baseline
  Assessed by stop drinking, increase (+50%), slight increase, decrease (-50%), slight decrease or no change of drinking after the start of pandemic
Covid-19 related drinking behavioral changes at 6-month | at 6-month
  Assessed by stop drinking, increase (+50%), slight increase, decrease (-50%), slight decrease or no change of drinking after the start of pandemic. The changes will be compared between the intervention group and control group at 6-month
Covid-19 related drinking behavioral changes at 12-month | at 12-month
  Assessed by stop drinking, increase (+50%), slight increase, decrease (-50%), slight decrease or no change of drinking after the start of pandemic. The changes will be compared between the intervention group and control group at 12-month

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Thomas GN, Wang MP, Ho SY, Mak KH, Cheng KK, Lam TH. Adverse lifestyle leads to an annual excess of 2 million deaths in China. PLoS One. 2014 Feb 26;9(2):e89650. doi: 10.1371/journal.pone.0089650. eCollection 2014. PMID 24586936
- [Background] Gore FM, Bloem PJ, Patton GC, Ferguson J, Joseph V, Coffey C, Sawyer SM, Mathers CD. Global burden of disease in young people aged 10-24 years: a systematic analysis. Lancet. 2011 Jun 18;377(9783):2093-102. doi: 10.1016/S0140-6736(11)60512-6. Epub 2011 Jun 7. PMID 21652063
- [Background] Wang MP, Ho SY, Lam TH. Underage alcohol drinking and medical services use in Hong Kong: a cross-sectional study. BMJ Open. 2013 May 28;3(5):e002740. doi: 10.1136/bmjopen-2013-002740. PMID 23793697
- [Background] Huang R, Ho SY, Wang MP, Lo WS, Lam TH. Reported alcohol drinking and mental health problems in Hong Kong Chinese adolescents. Drug Alcohol Depend. 2016 Jul 1;164:47-54. doi: 10.1016/j.drugalcdep.2016.04.028. Epub 2016 Apr 25. PMID 27177803
- [Background] Department of Health. Report of population health survey 2014/15, Hong Kong SAR; 2018. Retrived at 24 Oct 2018 from: https://www.chp.gov.hk/en/static/51256.html
- [Background] Kaner EF, Beyer FR, Muirhead C, Campbell F, Pienaar ED, Bertholet N, Daeppen JB, Saunders JB, Burnand B. Effectiveness of brief alcohol interventions in primary care populations. Cochrane Database Syst Rev. 2018 Feb 24;2(2):CD004148. doi: 10.1002/14651858.CD004148.pub4. PMID 29476653
- [Background] Fachini A, Aliane PP, Martinez EZ, Furtado EF. Efficacy of brief alcohol screening intervention for college students (BASICS): a meta-analysis of randomized controlled trials. Subst Abuse Treat Prev Policy. 2012 Sep 12;7:40. doi: 10.1186/1747-597X-7-40. PMID 22967716
- [Background] Kaner EF, Beyer FR, Garnett C, Crane D, Brown J, Muirhead C, Redmore J, O'Donnell A, Newham JJ, de Vocht F, Hickman M, Brown H, Maniatopoulos G, Michie S. Personalised digital interventions for reducing hazardous and harmful alcohol consumption in community-dwelling populations. Cochrane Database Syst Rev. 2017 Sep 25;9(9):CD011479. doi: 10.1002/14651858.CD011479.pub2. PMID 28944453
- [Background] Larimer ME, Cronce JM, Lee CM, Kilmer JR. Brief intervention in college settings. Alcohol Res Health. 2004-2005;28(2):94-104. PMID 19006997
- [Background] Moyer A, Finney JW, Swearingen CE, Vergun P. Brief interventions for alcohol problems: a meta-analytic review of controlled investigations in treatment-seeking and non-treatment-seeking populations. Addiction. 2002 Mar;97(3):279-92. doi: 10.1046/j.1360-0443.2002.00018.x. PMID 11964101
- [Background] Fowler LA, Holt SL, Joshi D. Mobile technology-based interventions for adult users of alcohol: A systematic review of the literature. Addict Behav. 2016 Nov;62:25-34. doi: 10.1016/j.addbeh.2016.06.008. Epub 2016 Jun 7. PMID 27310031
- [Background] Kypri K, Hallett J, Howat P, McManus A, Maycock B, Bowe S, Horton NJ. Randomized controlled trial of proactive web-based alcohol screening and brief intervention for university students. Arch Intern Med. 2009 Sep 14;169(16):1508-14. doi: 10.1001/archinternmed.2009.249. PMID 19752409
- [Background] Kypri K, Vater T, Bowe SJ, Saunders JB, Cunningham JA, Horton NJ, McCambridge J. Web-based alcohol screening and brief intervention for university students: a randomized trial. JAMA. 2014 Mar 26;311(12):1218-24. doi: 10.1001/jama.2014.2138. PMID 24668103
- [Background] Hoermann S, McCabe KL, Milne DN, Calvo RA. Application of Synchronous Text-Based Dialogue Systems in Mental Health Interventions: Systematic Review. J Med Internet Res. 2017 Jul 21;19(8):e267. doi: 10.2196/jmir.7023. PMID 28784594
- [Background] Luk TT, Li WHC, Cheung DYT, Wong SW, Kwong ACS, Lai VWY, Chan SS, Lam TH, Wang MP. Chat-based instant messaging support combined with brief smoking cessation interventions for Chinese community smokers in Hong Kong: Rationale and study protocol for a pragmatic, cluster-randomized controlled trial. Contemp Clin Trials. 2019 Feb;77:70-75. doi: 10.1016/j.cct.2018.12.013. Epub 2018 Dec 26. PMID 30593882
- [Background] Bock BC, Barnett NP, Thind H, Rosen R, Walaska K, Traficante R, Foster R, Deutsch C, Fava JL, Scott-Sheldon LA. A text message intervention for alcohol risk reduction among community college students: TMAP. Addict Behav. 2016 Dec;63:107-13. doi: 10.1016/j.addbeh.2016.07.012. Epub 2016 Jul 18. PMID 27450909
- [Background] Michie S, Whittington C, Hamoudi Z, Zarnani F, Tober G, West R. Identification of behaviour change techniques to reduce excessive alcohol consumption. Addiction. 2012 Aug;107(8):1431-40. doi: 10.1111/j.1360-0443.2012.03845.x. Epub 2012 Apr 17. PMID 22340523
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Derived] Chau SL, Luk TT, Wong BYC, Wu YS, Cheung YTD, Ho SY, Kim JH, Lo HHM, Lam TH, Wang MP. A Brief Intervention With Instant Messaging or Regular Text Messaging Support in Reducing Alcohol Use: A Randomized Clinical Trial. JAMA Intern Med. 2024 Jun 1;184(6):641-649. doi: 10.1001/jamainternmed.2024.0343. PMID 38587827
- [Derived] Chau SL, Wong YC, Zeng YP, Lee JJ, Wang MP. Perceptions of Using Instant Messaging Apps for Alcohol Reduction Intervention Among University Student Drinkers: Semistructured Interview Study With Chinese University Students in Hong Kong. JMIR Form Res. 2023 Feb 27;7:e40207. doi: 10.2196/40207. PMID 36848207